CLINICAL TRIAL: NCT06755528
Title: Effect of Shockwaves on Fallopian Tubes Adhesion: a Randomized Controlled Trial
Brief Title: Effect of Shockwaves on Fallopian Tubes Adhesion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shorouk Fawzy Mohamed, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003490
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Fallopian Tube Adhesion
MeSH Terms: interventions — Chitosan; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical therapy group (Active Comparator): The participants will receive medical therapy for fallopian tube adhesions as prescribed by the gynecologist
  Interventions: Drug: Chitosan
- Medical therapy and Shockwave therapy group (Experimental): The participants will receive medical therapy plus shockwave therapy (1 session per week for 4 weeks).
  Interventions: Drug: Chitosan; Device: shockwave therapy

INTERVENTIONS:
Drug: Chitosan — The participants will receive medications for fallopian tube adhesions (Chitosan (glucosamine (GIcN) and N-acetylglucosamine (GIcNAc) units,1 tablet per day) as prescribed by the gynecologist
Device: shockwave therapy — The participants will receive shockwave with the following parameters: sonic pulses characterized by: high peak pressure, up to 100 mpa (500 bar) or even more, rapid rise in pressure (<10 ns), short duration (<10 μs) and a broad range of frequency. The energy flux density was 0.09 to 0.16 mJ/mm2; with a frequency of 5 Hz and 2000 impulses, i session per week for 4 weeks.
  Arms: Medical therapy and Shockwave therapy group

SUMMARY:
The purpose of this study is to determine the effect of shock waves on fallopian tube adhesions.

DETAILED DESCRIPTION:
Tubal factor infertility accounts for approximately 40% of the cases of female infertility. Identifiable causes of tubal infertility are post-infectious tubal damage, endometriosis-related adhesions, and postsurgical adhesion formation.

Although surgical management is considered as a common choice for treating blocked tubes or adhesion it has many complications such as: infection, creation of more scar tissue, damage to organs and bleeding.

Shock waves is a modality that exerts an anti-inflammatory action and regenerative effect as well biological model. Shock waves can be nowadays considered an effective, safe, versatile, repeatable, noninvasive therapy for the treatment of many musculo-skeletal diseases, and for some pathological conditions where regenerative effects are desirable, especially when some other noninvasive/conservative therapies have failed.

For these reasons and complications of surgery, This study aims to examine the effect of shockwaves therapy on fallopian tubes adhesion

ELIGIBILITY:
Inclusion Criteria:

* Their ages will be ranged from 25 to 35 years old.
* Their body mass index (BMI) will be less than 35kg/m².
* All women will be diagnosed with fallopian tubes adhesion by the physician.
* They have regular menstrual cycles.
* All Patients have secondary infertility and they have previous caesarean section).

Exclusion Criteria:

* Any gynecological diseases (uterine prolapse, retroversion flexion of the uterus or chronic pelvic pain).
* Leukemia or tumor (spinal or pelvic tumor).
* Diabetes mellitus, hypertension, heart diseases, cardiovascular diseases and skin diseases.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of Fallopian tube adhesions | 4 weeks
  Pelvic abdominal ultrasound (ultrasound scanning system, SN.w7c1882026) will be used to assess fallopian tube adhesions for all participants in both groups before and after the treatment protocol (4 weeks)
Detection of Fallopian tube patency | 4 weeks
  Hysterosalpingography (DMC GmbH, 22335 Hamburg): it is a radiologic procedure that will be used to assess fallopian tube patency ( if the fallopian tube is opened or not) for all women in both groups before and after the treatment protocol (4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Fekry, PHD, Study Director — Al-Agoza Police Hospital; Soheir El-kosery, Professor, Study Chair — Cairo University